CLINICAL TRIAL: NCT02160080
Title: Boceprevir Treatment in Liver Pre-transplant HCV Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hu Tsung-Hui (Other)
Responsible Party: Sponsor-Investigator, Hu Tsung-Hui, Tsung-Hui Hu MD.PhD, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB:102-4331A
Record Dates: First submitted 2014-04-11; First posted 2014-06-10 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Late Complication From Liver Transplant
Keywords: Boceprevir;; Liver pre-transplant
MeSH Terms: interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Boc+Peg-int alfa+Rbv (Experimental): Boceprevir 800mg/TID+Pegylated interferon alfa+Ribavirin
  Interventions: Drug: Boceprevir 800mg/TID+Pegylated interferon alfa+Ribavirin

INTERVENTIONS:
Drug: Boceprevir 800mg/TID+Pegylated interferon alfa+Ribavirin — Boceprevir 800mg/TID+Pegylated interferon alfa+Ribavirin
  Other Names: Victrelis (Boceprevir)

SUMMARY:
End-stage liver disease due to hepatitis C virus (HCV) is the most common indication for liver transplantation(LT) worldwide (30~40%). Within 5 years, about 25-30% of liver transplant recipients with recurrent hepatitis C would progress to liver cirrhosis (Ponziani et. Al, 2011), it also accounts for 2/3 of graft failure and deaths after liver transplantation.(Bzowej et al., 2011)

Kaohsiung Chang Gung Memorial Hospital continue to have at least 45 HCV-related liver disease patients awaiting for liver transplantation annually. If the HCV viral load can be significantly reduced or sustained virologic response (SVR) can be achieved by triple therapy with Pegylated interferon alfa(PEG)/Ribavirin(RBV)/Boceprevir(BOC) treatment before liver transplantation(LT), the graft re-infection of HCV can be prevented. By this way, we can reduce the risk of early fibrosis progression in the liver graft, and hopefully, improving graft and patient survival after liver transplantation.(Toniutto, 2008)(Ponziani et al, 2011).

We aim to conduct an prospective, open label, single arm study. This study design is single arm to treat HCV patients with Pegylated interferon alfa(PEG)/Ribavirin(RBV)/Boceprevir(BOC) triple therapies before liver transplantation for patients with detectable HCV RNA. The total number of patients would be around 20 cases included in the study and all of them will take Pegylated interferon alfa(PEG)/Ribavirin(RBV)/Boceprevir(BOC) triple therapy. The experimental regimen contains 4 week lead-in therapy with Peg-Interferon α-2b plus Ribavirin. Then after, triple therapy with Boceprevir + Peg-Interferon α-2b + Ribavirin will be used for at least 16 weeks or maximal 44 weeks before transplantation. Normal practice based on the treatment protocol of the Kaohsiung Chang Gung Memorial Hospital liver transplant center will be done before enrollment. Patients will be monitored for all the efficacy and safety endpoints during the treatment period. HCV RNA will be checked at time of transplant. Finally, patients will received regular monitoring of HCV RNA 1, 3, 6, 9, 12 months after liver transplantation.

DETAILED DESCRIPTION:
End-stage liver disease due to hepatitis C virus (HCV) is the most common indication for liver transplantation(LT) worldwide (30~40%). Within 5 years, about 25-30% of liver transplant recipients with recurrent hepatitis C would progress to liver cirrhosis (Ponziani et. Al, 2011), it also accounts for 2/3 of graft failure and deaths after liver transplantation.(Bzowej et al., 2011)

Kaohsiung Chang Gung Memorial Hospital continue to have at least 45 HCV-related liver disease patients awaiting for liver transplantation annually. If the HCV viral load can be significantly reduced or sustained virologic response (SVR) can be achieved by triple therapy with pegylated interferon alfa (PEG)/Ribavirin(RBV)/Boceprevir(BOC) treatment before liver transplantation(LT), the graft re-infection of HCV can be prevented. By this way, we can reduce the risk of early fibrosis progression in the liver graft, and hopefully, improving graft and patient survival after liver transplantation.(Toniutto, 2008)(Ponziani et al, 2011).

We aim to conduct a prospective, open label, single arm study. This study design is single arm to treat HCV patients with pegylated interferon alfa (PEG)/Ribavirin(RBV)/Boceprevir(BOC) triple therapies before liver transplantation for patients with detectable HCV RNA. The total number of patients would be around 20 cases included in the study and all of them will take pegylated interferon alfa (PEG)/Ribavirin(RBV)/Boceprevir(BOC) triple therapy. The experimental regimen contains 4 week lead-in therapy with Peg-Interferon α-2b plus Ribavirin, followed by Boceprevir + Peg-Interferon α-2b + Ribavirin for at least 16 weeks or maximal 44 weeks before transplantation. The treatment will be discontinued immediately at time of liver transplantation. Normal practice based on the treatment protocol of the Kaohsiung Chang Gung Memorial Hospital liver transplant center will be done before enrollment.

-Treatment Stopping Rules-

If the patient has HCV RNA >100 IU/ml at week 12 after the beginning of treatment with peg interferon plus ribavirin, i.e. 8 weeks after the initiation of therapy with boceprevir, all HCV medications are to be discontinued.

If the patient has detectable HCV RNA at Week 24 after the beginning of treatment with peg interferon plus ribavirin, i.e. 20 weeks after the initiation of therapy with boceprevir, all HCV medications are to be discontinued.

Monitoring of Patients during Treatment Complete blood counts should be obtained pretreatment, Treatment Week 4, Treatment Week 8, and thereafter, as clinically appropriate. If serum hemoglobin is <10 g/dL, a decrease in dosage of ribavirin and/or administration with erythropoietin (epoetin alfa) may be warranted.

-Primary Outcome Measure: Title: Number of Participants with Adverse Events as a Measure of Safety Time Frame: Up to the time of liver transplant

-Secondary Outcome Measures: Title: HCV-RNA (Hepatitis C virus RNA) level Time Frame: Baseline, Treatment Week 12 , Treatment Week 24. A follow-up test is recommended 24 weeks after the completion of treatment, or at time of liver transplant. Finally, patients will receive regular monitoring of HCV RNA 1, 3, 6, 9, 12 months after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 20 years and older
2. Chronic infection with genotype 1 hepatitis C virus proven with positive PCR
3. Liver cirrhosis while awaiting liver transplantation
4. Patient with compensated liver functions
5. With or without hepatocellular carcinoma.
6. Naive or experienced (failure) to HCV antiviral treatmentFailure is defined according to the following terminology:

   * Relapsing patient: HCV RNA undetectable at the end of treatment, becoming detectable again after the discontinuation of treatment
   * Breakthrough: increase of viremia of 1 log or more during the treatment
   * Non-responding patient with partial response: HCV RNA detectable at W24 without ever having been undetectable and with a decrease in HCV RNA ≥ 2 log at W12
   * Non-responding patient with null response: decrease in HCV RNA < 2 log at W12
7. No need for prior treatment wash-out
8. Written patient informed consent

Exclusion Criteria:

1. Non controlled sepsis
2. Platelets < 50,000/mm3
3. Neutrophil granulocyte levels < 1000/mm3
4. Creatinine clearance < 50 mL/min
5. Hb < 10 g/dL
6. Uncontrolled psychiatric problems
7. Hypersensitivity or contraindications to any component of boceprevir formulation
8. Contraindication to interferon or ribavirin
9. HIV coinfection
10. HBV coinfection (unless this is treated effectively with analogues, as proven by undetectable viremia for at least 12 months)
11. Other infectious disease underway
12. Neoplastic disease other than hepatocellular carcinoma during the previous year, or neoplastic disease for which the prognosis is less than 3 years
13. Treatment with immunosuppressors (including corticosteroids), antivirals other than those for the study, except aciclovir
14. Current or anticipated use of any of the following prohibited medications: midazolam, pimozide, amiodarone, flecainide, propafenone, quinidine, and ergot derivatives
15. Person participating in another study including an exclusion period that is still underway during pre-enrollment
16. Pregnancy, breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | within 1 year

SECONDARY OUTCOMES:
HCV-RNA (Hepatitis C virus RNA) level | within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hui Hu, Ph.D, Principal Investigator — Department of Internal Medicine
Locations (1):
- 123, Ta Pei Road, Niao Sung Hsiang, Kaohsiung Hsien, Taiwan